CLINICAL TRIAL: NCT03319758
Title: Esthetic, Clinical and Patient-centered Outcomes Following Immediate Implant Placement With Thin or Dehiscence Buccal Bone Wall in the Anterior Maxilla
Brief Title: Esthetic and Radiographic Outcomes Following Immediate Implant Placement With Thin or Dehiscence Buccal Bone Wall
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Baoxin Huang, Principal Investigator, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Baoxin Huang
Record Dates: First submitted 2017-09-14; First posted 2017-10-24 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Jaw, Edentulous, Partially; Acquired Absence of Single Tooth
Keywords: bone augmentation; esthetics; immediate implant; buccal bone defects
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- thin or dehiscences buccal plate (Experimental): Immediate implant placement used bone augmentation in combination with an absorbable collagen membrane with thin or dehiscences buccal plate.
  Interventions: Procedure: buccal bone augmentation

INTERVENTIONS:
Procedure: buccal bone augmentation — Subjects in need of one implant replacing tooth to be removed in the maxilla within region 13-23 are included. At least 15 patients are recruited.

SUMMARY:
The aim of this prospective study was to evaluate the soft and hard tissue changes of immediate implant placement with buccal bone augmentation in sites with thin labial bone wall in the anterior maxillary zone.

DETAILED DESCRIPTION:
The objective of this prospective controlled clinical trial is to compare the esthetic and radiographic outcomes following immediate implant placement with thin or dehiscences buccal plate using bone augmentation in combination with an absorbable collagen membrane. Subjects in need of one implant replacing tooth to be removed in the maxilla within region 13-23 are included. At least 15 patients are recruited. No implant-supported temporary restorations are used during the first 4 months. After a screw-retained provisional phase of 2 months, a ﬁnal impression is taken at implant level and take-in definitive crown. Patients are recalled for oral hygiene maintenance and prosthetic controls every 6 months for the entire duration of the study.

ELIGIBILITY:
The inclusion criteria were as follows:

1. 18 to 70-year-old;
2. Stable periodontal and systemic health (American Society of Anesthesiologists classification I or II);
3. Single maxillary anterior teeth (canine to canine);
4. Bone thickness less than 1mm at 4mm apical to cementum-enamel junction (CEJ-4)；
5. Presence of adjacent nature tooth;
6. Good compliance;
7. No palatal vertical bone loss;
8. Good oral hygiene.

Exclusion criteria are as follow:

1. Uncontrolled periodontal or systemic disease;
2. General psychiatric contraindications;
3. More than 20 cigarettes per day;
4. History of head and neck radiotherapy；
5. Pregnant or expecting to be pregnant;
6. Patients with local or generalized healing limitations;
7. Bruxism or other destructive parafunctional habits;
8. Drug abuse or alcohol abuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Radiographic bone volume | Up to 10 years after baseline
  Radiographic bone volume be assessed at pre-operation, 0 ,0.5, 1, 1.5, 3.5, 5.5, 7.5, 10.5 years after implant placement.

SECONDARY OUTCOMES:
Change of Pink and white esthetic scores (PES/WES) | Change from baseline up to 10 years after implantation
  Baseline will be at the time of implant placement.Pink and white esthetic scores (PES/WES) will be recorded at 0.5, 1.5, 3.5, 5.5, 7.5, 10.5 years after implant placement.
Visual analogue scale (VAS) | Up to 10 years after baseline
  A questionnaire will be recorded at pre-operation, 0.5, 1, 1.5, 3.5, 5.5, 7.5, 10.5 years after implant placement
Oral health impact profile shortened version (OHIP-I) | Up to 10 years after baseline
  A questionnaire will be recorded at pre-operation, 0.5, 1, 1.5, 3.5, 5.5, 7.5, 10.5 years after implant placement.
Buccal marginal recession | Up to 10 years after baseline
  Buccal marginal recession will be assessed at pre-operation, 0.5, 1, 1.5, 3.5, 5.5, 7.5, 10.5 years after implant placement.
Papilla volume | Up to 10 years after baseline
  Papilla volume will be assessed at 0.5, 1, 1.5, 3.5, 5.5, 7.5, 10.5 years after implant placement.
Width of keratinized gingiva | Up to 10 years after baseline
  Width of keratinized gingiva will be assessed at 0.5, 1, 1.5, 3.5, 5.5, 7.5, 10.5 years after implant placement.
Implant survival | Up to 10 years after baseline
  Implant survival will be assessed at 0.5, 1, 1.5, 3.5, 5.5, 7.5, 10.5 years after implant placement.
Probing depth | Up to 10 years after baseline
  Probing depth will be assessed at pre-operation, 0.5, 1, 1.5, 3.5, 5.5, 7.5, 10.5 years after implant placement.
Modified plaque index | Up to 10 years after baseline
  Modified plaque index will be assessed at pre-operation, 0.5, 1, 1.5, 3.5, 5.5, 7.5, 10.5 years after implant placement.
Modified bleeding index | Up to 10 years after baseline
  Modified bleeding index will be assessed at pre-operation, 0.5, 1, 1.5, 3.5, 5.5, 7.5, 10.5 years after implant placement.

CONTACTS AND LOCATIONS:
Overall Officials: Baoxin Huang, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Guanghua School of Stomatology,Hospital of Stomatology,Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sarnachiaro GO, Chu SJ, Sarnachiaro E, Gotta SL, Tarnow DP. Immediate Implant Placement into Extraction Sockets with Labial Plate Dehiscence Defects: A Clinical Case Series. Clin Implant Dent Relat Res. 2016 Aug;18(4):821-9. doi: 10.1111/cid.12347. Epub 2015 Apr 27. PMID 25916859
- [Result] Barone A, Ricci M, Romanos GE, Tonelli P, Alfonsi F, Covani U. Buccal bone deficiency in fresh extraction sockets: a prospective single cohort study. Clin Oral Implants Res. 2015 Jul;26(7):823-30. doi: 10.1111/clr.12369. Epub 2014 Mar 31. PMID 24684275
- [Result] Aloy-Prosper A, Penarrocha-Oltra D, Penarrocha-Diago M, Penarrocha-Diago M. Dental implants with versus without peri-implant bone defects treated with guided bone regeneration. J Clin Exp Dent. 2015 Jul 1;7(3):e361-8. doi: 10.4317/jced.52292. eCollection 2015 Jul. PMID 26330931